CLINICAL TRIAL: NCT00770237
Title: Effects of Smoking Cues on Tobacco Craving Responses and the Reinforcing Efficacy of Cigarettes in Smokers With and Without Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, MPRC, Deanna L. Kelly, Pharm.D., BCPP, University of Maryland, Baltimore
Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: HP-00042356; NIDA 430
Record Dates: First submitted 2008-10-07; First posted 2008-10-09 (Estimated); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Schizophrenia; Nicotine Dependence
Keywords: Smoking; Nicotine; Schizophrenia
MeSH Terms: conditions — Schizophrenia; Tobacco Use Disorder; Smoking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cues (Experimental): Outcome Measures During cue trials, primary measures include craving (TCQ-SF, VAS), mood (mood form, VAS), and autonomic (heart rate, blood pressure, skin conductance and temperature) responsivity. During self-administration trials, primary measures include breakpoint (final ratio completed), total number of responses, and number of cigarette puffs earned and taken. Secondary measures include baseline smoking history, mood form, TCQ-SF, CO, FTND, and urinary cotinine and 3-hydroxycotinine (3-HC).
  Interventions: Behavioral: Smoking Cues; Behavioral: Neutral Cues

INTERVENTIONS:
Behavioral: Smoking Cues — In the smoking cue condition, a pack of the participants preferred brand of cigarettes, a lighter, and an ashtray will be under the tray cover. In the neutral cue condition, a pack of unsharpened pencils, a pencil sharpener, and a small notepad will be under the cover. When instructed, the participant will lift the cover on the tray. In the smoking cue condition, participants will take one cigarette out of the pack, light it without puffing, hold it for 1 minute, extinguish the cigarette, and replace the cover on the tray.
Behavioral: Neutral Cues — In the neutral cue condition, participants will take one pencil out of the pack, sharpen it, hold it for 1 minute as if to write on the notepad, and then replace the cover. Participants will complete the VAS during cue exposure and the TCQ-SF, VAS, and mood form immediately and 15 minutes after cue presentation; physiological measures will be recorded continuously.

SUMMARY:
In this study, we will compare cue-reactivity in smokers with and without schizophrenia and the influence of smoking cues on responding for cigarette puffs under a PR schedule of reinforcement. Given the high prevalence of smoking among individuals with schizophrenia, understanding some of the environmental factors that serve to maintain nicotine dependence is a critical step in improving smoking cessation treatment outcomes. Establishing and validating a laboratory model of cue-elicited responsivity and cigarette self- administration will allow the investigation of the efficacy of anti-craving medications in people with schizophrenia.

Specific Aims 1) To compare the effects of smoking versus neutral cues on craving, mood, and autonomic responsivity in smokers with schizophrenia and smokers without schizophrenia. 2) To compare the effects of smoking versus neutral cues on the reinforcing efficacy of tobacco cigarettes in smokers with schizophrenia and smokers without schizophrenia.

Outcome Measures During cue trials, primary measures include craving (TCQ-SF, VAS), mood (mood form, VAS), and autonomic (heart rate, blood pressure, skin conductance and temperature) responsivity. During self-administration trials, primary measures include breakpoint (final ratio completed), total number of responses, and number of cigarette puffs earned and taken. Secondary measures include baseline smoking history, mood form, TCQ-SF, CO, FTND, and urinary cotinine and 3-hydroxycotinine (3-HC).

The ratio of 3-HC/cotinine is a phenotypic biomarker of the rate of nicotine metabolism, which has been shown to be associated with level of nicotine dependence, various smoking behaviors, and treatment outcome (Ho & Tyndale, 2007). We will correlate the primary measures with the 3-HC/cotinine ratio to explore possible relationships for future study.

ELIGIBILITY:
* Inclusion Criteria for Schizophrenia Patients

  1. 18-64 year old males and females
  2. Smoking at least 10 cigarettes per day for at least 1 year
  3. Urinary cotinine level ≥ 100 ng/ml (NicAlert® reading ≥ 3)
  4. Current DSM-IV diagnosis of schizophrenia and stable medication regimen (see above)
  5. Medically healthy as determined by screening criteria
* Inclusion Criteria for Healthy Volunteers

  1. 18-64 year old males and females
  2. Smoking at least 10 cigarettes per day for at least 1 year
  3. Urinary cotinine level ≥ 100 ng/ml (NicAlert® reading ≥ 3)
  4. Medically and psychologically healthy as determined by screening criteria
* Exclusion Criteria for Schizophrenia Patients

  1. Current interest in reducing or quitting tobacco use
  2. Treatment for tobacco dependence in the past 3 months
  3. Use of nicotine replacement products, bupropion, or varenicline in the past 3 months
  4. Consumption of more than 15 alcoholic drinks per week during the past month
  5. Use of any illicit drug more than twice per week during the past month
  6. Current use of any medication that would interfere with the protocol in the opinion of MAI (e.g., medications that would interfere with the cue reactivity portion of the study including, but not limited to, antidepressants, first-generation antipsychotics, and mood stabilizers)
  7. Under the influence of a drug or alcohol at experimental sessions
  8. Pregnant, nursing, or become pregnant during the study
* Exclusion Criteria for Healthy Volunteers

  1. Current interest in reducing or quitting tobacco use
  2. Treatment for tobacco dependence in the past 3 months
  3. Use of nicotine replacement products, bupropion, or varenicline in the past 3 months
  4. Consumption of more than 15 alcoholic drinks per week during the past month
  5. Use of any illicit drug more than twice per week during the past month
  6. Current use of any medication that would interfere with the protocol in the opinion of MAI (e.g., medications that would interfere with the cue reactivity portion of the study including, but not limited to, antidepressants, antipsychotics, and mood stabilizers)
  7. Under the influence of a drug or alcohol at experimental sessions
  8. Pregnant, nursing, or become pregnant during the study

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2008-10 (Actual); Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To compare the effects of smoking versus neutral cues on craving, mood, and autonomic responsivity in smokers with schizophrenia and smokers without schizophrenia. | 7-10 Days

CONTACTS AND LOCATIONS:
Overall Officials: Deanna L Kelly, Pharm.D, BCPP, Principal Investigator — University of Maryland, College Park; Stephen J Heishman, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- Maryland Psychiatric Research Center (MPRC) Outpatient Research Program (ORP); the MPRC Treatment Research Program (TRP), Catonsville, Maryland, United States